CLINICAL TRIAL: NCT04988620
Title: Cold Stored Whole Blood in Treatment of Bleeding in Patients Undergoing Cardiothoracic Surgery
Brief Title: Cold Stored Whole Blood in Cardiothoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/01294
Record Dates: First submitted 2021-06-04; First posted 2021-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Exchange Transfusion, Whole Blood

STUDY DESIGN:
Intervention Model Description: Test group ( Whole Blood stored for 15-21 days) versus Control group(s) (Whole Blood stored for less than 7 days, Whole Blood stored for 8-14 days and/or Standard Blood Component treatment)
Who Masked: Participant, Care Provider
Masking Description: The participant and clinical personell ordering and evalutaing the effect of transfusion will be blinded, so will also the investigators performing the statistical evaluation of the results. The project co-workers preparing the whole blood units and perforing laboratory analysis will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Whole Blood stored for 15-21 days (Experimental): CPD Whole Blood leukoreduced with a platelet-sparing filter and stored cold for 15-21 days
  Interventions: Other: Whole Blood transfusion
- Whole Blood stored for less than 7 days (Active Comparator): CPD Whole Blood leukoreduced with a platelet-sparing filter and stored cold for less than 7 days. We aim at using as fresh as possible.
  Interventions: Other: Whole Blood transfusion
- Whole Blood stored for 8-14 days (Active Comparator): CPD Whole Blood leukoreduced with a platelet-sparing filter and stored cold for 8-14 days. This group may be added if deemed of interest after interim analysis.
  Interventions: Other: Whole Blood transfusion
- Standard Blood Component (Active Comparator): This group may be added for comparison if deemed of interest after interim analysis.
  Interventions: Other: Whole Blood transfusion

INTERVENTIONS:
Other: Whole Blood transfusion — In this study the effect of storage time of whole blood will be investigated. Intervention is storage of whole blood.

SUMMARY:
In vitro platelet function and post-transfusion platelet recovery of platelets stored in whole blood decline during storage. In this pilot randomized clinical trial we aim to investigate the impact of storage time of whole blood on the effect and safety in treatment of immediate blood loss in patients undergoing complex cardiothoracic surgery. The study is designed as an exploratory superiority study to support feasibility and provide critical guidance for future, more definitive randomized trials. In the study the test group will receive CPD whole blood leukocyte-depleted with a platelet-sparing filter and stored for 15-21 days whereas the control group patients will receive leukocyte-depleted CPD whole blood stored for less than 7 days.

DETAILED DESCRIPTION:
A challenge for implementation of Whole Blood programs in civilian health services has been an uncertainty regarding the impact of storage on the clinical effect of the whole blood transfusion, especially when it comes to platelet function which is essential to hemostasis. In vitro platelet function and post-transfusion platelet recovery decline with increasing storage time of the whole blood.

In this pilot randomized clinical trial we aim to investigate the impact of storage time of whole blood on the effect and safety in treatment of immediate blood loss in patients undergoing complex cardiothoracic surgery. The study is designed as an exploratory superiority study to support feasibility and provide critical guidance for future, more definitive randomized trials. In the study the test group will receive CPD whole blood leukocyte-depleted with a platelet-sparing filter and stored for 15-21 days whereas the control group patients will receive leukocyte-depleted CPD whole blood stored for less than 7 days. A control group receiving standard care (blood component-based transfusion) may be included.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing cardiothoracic, cardiac, or aortic surgery
2. Patients with complex surgical procedures and expected cardiopulmonary bypass (CPB) time over 120 minutes
3. Patients capable of providing informed consent to participate in the study

Exclusion Criteria:

1. Patients not capable of providing informed consent to participate or who will not provide informed consent
2. Patients with known congenital coagulopathies or hemostatic disorders (von Willebrands Disease, hemophilia etc)
3. Patients with known erythrocyte- or platelet/HLA antibodies
4. Patients with a particular increased surgical risk with expected need of ECMO
5. Patients with preoperative EuroScore II ≥ 30

5. RhD negative patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood loss | 24 hours (8:00 am morning after surgery)
  Comparison of postoperative immediate blood loss (measured by chest drain output and/or bleeding score) in patients receiving fresher or older cold stored whole blood.
Blood usage | 24 hours (8:00 am morning after surgery)
  Comparison of amount of whole blood and blood components given

SECONDARY OUTCOMES:
INR | 24 hours (8:00 am morning after surgery)
  Coagulation measured as INR
APTT | 24 hours (8:00 am morning after surgery)
  Coagulation measured as APTT
Thromboelastography | 24 hours (8:00 am morning after surgery)
  Thromboelastography (TEG6s)
Platelet aggregometry | 24 hours (8:00 am morning after surgery)
  Platelet aggregation measured by Multiplate impedance aggregometry (Mulitplate analyzer)
Platelet count | 24 hours (8:00 am morning after surgery)
  Platelet count
Hemoglobin concentration | 24 hours (8:00 am morning after surgery)
  Hemoglobin concentration
Erythrocyte count | 24 hours (8:00 am morning after surgery)
  Erythrocyte count
Hematocrit | 24 hours (8:00 am morning after surgery)
  Hematocrit or erytrocyte volume fraction, i.e.the volume percentage (vol%) of red blood cells (RBC) in blood,
Fibrinogen concentration | 24 hours (8:00 am morning after surgery)
  Fibrinogen concentration
Metabolomic profile | 24 hours (8:00 am morning after surgery)
  Investigation of blood cell metabolism and metabolic profile by use of high resolution mass spectometry
White blood cell count | 24 hours (8:00 am morning after surgery)
  White blood cell count
Bilirubin | Up to 7 days
  Hemolysis measured as Bilirubin
Haptoglobin | Up to 7 days
  Hemolysis measured as Haptoglobin
Lactate dehydrogenase | Up to 7 days
  Lactate dehydrogenase (LD)
Direct antiglobin test | Up to 7 days
  Direct antiglobin test (DAT)
Anti-A antibodies | Up to 7 days
  Anti-A antibodies
Anti-B antibodies | Up to 7 days
  Anti-B antibodies
Hemostatic agents | 24 hours (8:00 am morning after surgery)
  Use of hemostatic agents (coagulation factor concentrates, fibriongen concentrate)
Other medications | 24 hours (8:00 am morning after surgery)
  Use of other medications potentially affecting bleeding (including tranexamacid, calcium etc.)
Adverse events | 30 days
  Adverse events
Length of stay | 30 days
  Length of stay
Mortality | 30 days
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Einar K Kristoffersen, PhD, Study Chair — Helse Bergen
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No